CLINICAL TRIAL: NCT05658406
Title: Supplemental Perioperative Intravenous Crystalloids for Postoperative Nausea and Vomiting in Children Undergoing Oncological Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0305737
Record Dates: First submitted 2022-12-12; First posted 2022-12-20 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-09

CONDITIONS: Nausea and Vomiting, Postoperative
Keywords: Postoperative nausea and vomiting, oncological surgery
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Vomiting | interventions — Ringer's Lactate; Saline Solution

STUDY DESIGN:
Intervention Model Description: Patients will be prospectively and randomly assigned to one of the four groups (25 in each group). Random sequence generation and allocation concealment will be done using Computer-generated randomization. Supplemental crystalloid administration started after induction of anaesthesia (intraoperatively), in addition to standard fluid management. Patients will be divided into 4 groups:
  1. Group A: intraoperative infusion of 15 mL/kg/hour Ringer's lactate.
  2. Group B: intraoperative infusion of 10 mL/kg/hour Ringer's lactate.
  3. Group C: intraoperative infusion of 6 mL/kg/hour Ringer's lactate.
  4. Group D: standard fluid management alone.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Active Comparator): intraoperative infusion of 15 mL/kg/hour Ringer's lactate.
  Interventions: Drug: Ringer's Lactate
- Group B (Active Comparator): intraoperative infusion of 10 mL/kg/hour Ringer's lactate
  Interventions: Drug: Ringer's Lactate
- Group C (Active Comparator): intraoperative infusion of 6 mL/kg/hour Ringer's lactate.
  Interventions: Drug: Ringer's Lactate
- Group D (Placebo Comparator): standard fluid management alone
  Interventions: Drug: normal Saline

INTERVENTIONS:
Drug: Ringer's Lactate — infusion of 15 mL/kg/hour Ringer's lactate intraoperative
  Arms: Group A
Drug: Ringer's Lactate — infusion of 10 mL/kg/hour Ringer's lactate intraoperative .
  Arms: Group B
Drug: Ringer's Lactate — infusion of 6 mL/kg/hour Ringer's lactate intraoperative .
  Arms: Group C
Drug: normal Saline — standard fluid management: 4 ml for 1st 10 kg, 2 ml for the next 10 kg , 1 ml rest of body weight
  Arms: Group D

SUMMARY:
Postoperative nausea and vomiting (PONV) is a common complication in the paediatric population and is a source of significant morbidity. The incidence of PONV in children is alarmingly high, as it is estimated to be between 33.2% to 82% depending on patient risk factors. Even with the administration of prophylactic antiemetic medications, the risk of PONV can still be approximately 30%. Various independent risk factors have been implicated in the development of paediatric PONV. The following risk factors were identified: a duration of surgery 30 minutes or longer, age 3 years or older, strabismus, adenoidectomy, and tonsillectomy surgeries, a history of PONV in the child or immediate relatives (parents or siblings), use of volatile anaesthetic, use of opioids, increased postoperative pain, prolonged preoperative fast, and state of dehydration Significant improvement in patient satisfaction can be achieved if the incidence of PONV is decreased. Although not usually life-threatening, PONV may lead to complications commonly associated with vomiting, including dehydration, electrolyte imbalance, and aspiration of gastric contents. In some surgical cases, PONV has also led to wound complications, oesophageal rupture, subcutaneous emphysema, pneumomediastinum, and bilateral pneumothorax. PONV typically describes nausea, vomiting, or retching that can occur starting in the post-anaesthesia care unit (PACU) and continuing through the 24 hours following surgery. PONV occurs twice as often in children than in adults and can lead to longer PACU stays, delays in hospital discharge and subsequent unplanned readmissions, which ultimately lead to significant financial burden on the patients.

A variety of antiemetic regimens are recommended for the prevention and treatment of PONV in children, including pharmacotherapy with dexamethasone, 5HT-3 receptor antagonists, butyrophenones, prokinetics, anticholinergics and antihistamines.

Hydration is yet another important factor in the development of PONV in paediatric patients. Administration of intravenous dextrose-containing solutions may also prevent PONV. Investigation of the effect of perioperative intravenous crystalloid administration on PONV was initially motivated by the results of observational studies suggesting that perioperative volume status influenced postoperative complication rates. This work showed that PONV was among the most prevalent events after surgery and motivated subsequent inquiry into the relationship between perioperative volume resuscitation and PONV .

Multiple reviews have explained the complex physiology of nausea and vomiting. Briefly, the vomiting centre, located in the lateral reticular formation of the medulla, co-ordinates efferent activity to the respiratory, gastrointestinal, and abdominal musculature to produce vomiting. This centre receives afferent stimuli from a variety of sites: the pharynx, gastrointestinal tract chemo- and stretch receptors, the brain (including vestibular information from cranial nerve VIII), aortic baroreceptors, and the chemoreceptor trigger zone. The chemoreceptor trigger zone is a neural centre physiologically outside of the blood-brain barrier, which provides afferent information to the vomiting centre in response to noxious stimuli in the blood.

Patients particularly paediatrics typically present for surgery with a fluid deficit secondary to fasting, bleeding, bowel preparation, and other causes of dehydration. It has been proposed that brainstem, vestibular, and intestinal hypoperfusion, with concomitant ischaemia, may mediate nausea and vomiting. Supplemental intravenous crystalloids could serve to mitigate this effect; however, no proven explanation for the putative role of volume status in this model exists. Hypovolemia has been associated with a rise in postoperative morbidity and mortality ranging from PONV to other complications such as organ dysfunction . Hypovolemia from overnight fasting without adequate fluid replacement can cause adverse effects postoperatively . Intravenous crystalloids are widely administered before, during, and after procedures requiring general anaesthesia. They are inexpensive and have relatively few adverse effects. A prior systematic review has suggested that supplemental intravenous crystalloids may be effective in preventing PONV . However, studies of supplemental perioperative intravenous crystalloids were noted to vary widely on the specific volumes administered.

Despite evidence-based, multimodal prophylactic regimens, PONV remains a prevalent clinical problem . The use of pharmacologic agents alone reduces the risk of PONV but increases the risk of side effects. Intravenous crystalloids are an attractive treatment modality. Many different intravenous fluid interventions have been tested in a wide variety of surgical and anaesthetic contexts.

DETAILED DESCRIPTION:
The aim of this study is to test the hypothesis that intraoperative supplemental intravenous crystalloid fluid administration will reduce the incidence of postoperative nausea and vomiting in paediatric patients undergoing oncological surgical procedures under general anaesthesia.

Outcomes:

Primary outcomes:

We will analyse the risk of PONV occurring at different postoperative time points postoperatively (i.e., early, late). The early postoperative period will be defined as the period within six hours after surgery, while the late postoperative period will be defined as the time nearest to 24 hours after surgery. PON was defined as an unpleasant sensation associated with the urge to vomit. POV was defined as an attempted expulsion of gastric contents (vomiting or retching). PONV was defined as any nausea, vomiting, or both.

Secondary outcomes:

1. Risk of requiring antiemetic rescue medication during the postoperative period. Antiemetic rescue medication was defined as any additional intervention provided for the treatment of established PON, POV, or PON.
2. Risk of suffering a serious adverse event (any of: admission to high-dependency unit, postoperative cardiac or respiratory complication, or death).
3. To comprehensively determine the predictors of PONV as the dependant variable with age, gender, weight, operative time, treatment group, pain, fever, and preoperative chemotherapy as independent variables.

Patients and methods

This double-blind, prospective randomized controlled trial will be conducted in Borg Al-Arab Children's Cancer Centre, Alexandria University Hospitals in Borg Al-Arab, Alexandria, Egypt. After obtaining ethical committee approval and informed consent, we will study 100 patients, aged 3-13 years, with a diagnosis of malignancy, undergoing surgery. Parents will be given the option to give their children clear fluids up to 4 hours prior their arrival to the operating room. Screened participants will be excluded if:

1. They personally had a history of PONV or motion sickness;
2. A sibling or parent or both, had a history of PONV.
3. They received antiemetic medication in the 24 hours preceding surgery.
4. Their BMI exceeded 30 kg/m2.
5. They had a history of cardiovascular or renal disease.
6. Developmental delay or mental retardation, or both.
7. They significant intraoperative blood loss (> 30% blood volume loss).
8. They had a history of cardiorespiratory disease.
9. They had a history of renal or hepatic diseases.

Patients will be prospectively and randomly assigned to one of the four groups (25 in each group). Random sequence generation and allocation concealment will be done using Computer-generated randomization. Supplemental crystalloid administration started after induction of anaesthesia (intraoperatively), in addition to standard fluid management. Patients will be divided into 4 groups:

1. Group A: intraoperative infusion of 15 mL/kg/hour Ringer's lactate.
2. Group B: intraoperative infusion of 10 mL/kg/hour Ringer's lactate.
3. Group C: intraoperative infusion of 6 mL/kg/hour Ringer's lactate.
4. Group D: standard fluid management alone.

Perioperative management:

All children will be given midazolam at 0.5 mg/kg orally for sedation 30 min in preoperative holding area. Anaesthesia will induced with sevoflurane in oxygen. After induction a peripheral IV cannula will be inserted for intravenous access; none of the patients will receive any prophylactic antiemetic drugs. Anaesthesia will be maintained with endotracheal tube (ETT), and controlled ventilation using atracurium, sevoflurane, and oxygen. Anaesthesia will be supplemented with fentanyl 1 µg/kg during induction and a suitable regional analgesia technique for surgery. Monitoring will include electrocardiogram, blood pressure, endtidal CO2, temperature and pulse oximetry. The ETT Will be removed at the conclusion of surgery under a deep plane of anaesthesia.

Postoperative care will be standardized. Rescue antiemetics will be administered to patients if they were severely nauseated or vomited on more than one occasion using ondansetron 1-2 mg i.v., analgesia will be given to children complaining of pain using a pain scale monitoring for toddlers and young children. This will be consisted of oral analgesia (paracetamol). Perioperatively, the study investigators and postanesthesia care unit (PACU) nurses will be blinded to the allocation of the groups and the amount of fluid the subjects received.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of malignancy and undergoing surgery

Exclusion Criteria:

* They personally had a history of PONV or motion sickness;
* A sibling or parent or both, had a history of PONV.
* They received antiemetic medication in the 24 hours preceding surgery.
* Their BMI exceeded 30 kg/m2.
* They had a history of cardiovascular or renal disease.
* Developmental delay or mental retardation, or both.
* They significant intraoperative blood loss (> 30% blood volume loss)

Ages: 3 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2022-09-27 (Actual)

PRIMARY OUTCOMES:
risk of early postoperative nausea and vomiting | six hours after surgery
  The early postoperative period will be defined as the period within six hours after surgery,
risk of late postoperative nausea and vomiting | 24 hours after surgery
  late postoperative period will be defined as the time nearest to 24 hours after surgery

SECONDARY OUTCOMES:
Risk of requiring anti-emetic rescue medication | 24 hours after surgery.
  need for postoperative anti-emetic rescue medication.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria University Faculty of Medicin, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No